CLINICAL TRIAL: NCT02500199
Title: A Two-part Phase I, Open Label, Dose Escalation Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Pyrotinib in Patients With HER2-positive Solid Tumors Whose Disease Progressed on Prior HER2 Targeted Therapy
Brief Title: Phase I Study of Pyrotinib in Patients With HER2-positive Solid Tumors
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Hengrui Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SHRUS 1001
Record Dates: First submitted 2015-07-02; First posted 2015-07-16 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Breast Cancer; Gastric Cancer; Solid Tumors; NSCLC
Keywords: HER2 positive
MeSH Terms: conditions — Breast Neoplasms; Stomach Neoplasms | interventions — pyrotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Pyrotinib (Experimental): A two-part Phase I, open-label, dose escalation study to evaluate the safety, tolerability and pharmacokinetics of pyrotinib in patients with HER2-positive solid tumors whose disease progressed on prior HER2 targeted therapy
  Interventions: Drug: Pyrotinib

INTERVENTIONS:
Drug: Pyrotinib — Pyrotinib maleate, is provided as yellow, film-coated, immediate release tablets containing pyrotinib maleate at dosage strengths of 80 and 160 mg. Multiple tablets of pyrotinib will be administered daily to achieve targeted doses of pyrotinib: 320 mg, 400 mg, 480 mg, 560 mg and 640 mg. Tablets will be orally administered with water, once daily, 30 min after a meal.
  Other Names: SHR1258

SUMMARY:
Part 1: to assess the safety and tolerability of pyrotinib and to define the maximum tolerated dose (MTD) of pyrotinib in patients with Human Epidermal Growth Factor Receptor 2 (HER2)-positive advanced solid tumors (metastatic breast cancer, gastric cancer, or other solid tumors that have no targeted agent as standard of care).

Part 2: to estimate the overall response rate (ORR) for patients with HER2-positive metastatic breast cancer (mBC) and HER2 mutant non-small cell lung cancer (NSCLC) treated at the RP2D (or MTD).

DETAILED DESCRIPTION:
This is an open-label, dose escalation study of repeated doses of pyrotinib in patients with HER2-positive advanced solid tumors, including breast cancer, non small cell lung cancer.

Part 1 of the trial is dose escalation and is designed to enroll 3 to 6 patients in each dose group. Adverse events (AEs) will be assessed and monitored throughout the study. Dose-limiting toxicities (DLT) will be assessed from the first dose of study drug through day 28 in the first cycle of treatment.

Part 2 of the trial will consist of two independent arms: arm A for HER2 positive mBC and arm B for NSCLC with documented HER2 mutation will be investigated to further evaluate safety and the preliminary effectiveness and clinical benefits of pyrotinib as a single agent.

ELIGIBILITY:
The study is open to all males and females who meet the following inclusion criteria at screening and baseline to participate in the study.

To be included to participate in this study each patient must:

* be ≥ 18 years of age;
* have an Eastern Cooperative Oncology Group performance status of 0-1 (not declining within past 2 weeks, see Appendix 1);
* have confirmed HER2 gene amplified tumor fluorescence in-situ hybridization (FISH, HER2/cep17 ratio > 2) or HER2 overexpression (IHC 3+) or documented HER2 gene mutation. Documentation of HER2 status using FDA approved test(s) for HER2 testing specific for HER2 breast and gastric cancer is required prior to screening;
* for part 1:

  1. Patients with HER2 positive (defined as documented overexpression or amplification or mutation) metastatic breast cancer who have experienced disease progression following at least 2 prior anti-HER2 therapies for metastatic disease that contain trastuzumab with or without pertuzumab, prior T-DM1, or lapatinib therapy is required;
  2. Patients with HER2 positive metastatic gastric cancer who have disease progression on prior trastuzumab therapy;
  3. other HER2-positive solid tumors (defined as documented overexpression or amplification or mutation) that have no approved targeted agent as standard of care
* for part 2:

  1. Patients with HER2 positive metastatic breast cancer who have experienced disease progression after at least 2 prior anti-HER2 therapies for metastatic disease that contain trastuzumab with or without pertuzumab, prior T-DM1, or lapatinib therapy is required;
  2. Patients with documented HER2 mutated NSCLC whose disease progressed on prior therapy;
  3. Patients in Part 2 extension must have at least one measurable lesion as defined by modified Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 criteria;
* Left ventricular ejection fraction within institutional limits of normal (by multi gated acquisition scan or echocardiography;
* have the required screening laboratory values including the following parameters:

  1. Absolute neutrophil count ≥ 1.5×109/L (1,500/mm3);
  2. Platelets ≥ 75×109/L (75,000/mm3);
  3. Hemoglobin ≥ 9.0 g/dL (90 g/L);
  4. Total bilirubin ≤ 1.5× upper limit of normal (ULN);
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN; for patients with liver metastases, ALT and AST ≤ 5×ULN;
  6. Serum creatinine ≤ 1.5×ULN;
* have a life expectancy of > 12 weeks;
* for female patients who are of child bearing potential, a negative serum pregnancy test result before study entry. A female patient of childbearing potential is one who is biologically capable of becoming pregnant. This includes women who are using contraceptives or other means of birth control or whose sexual partners are either sterile or using contraceptives;
* and who have provided informed consent by signing the informed consent form.

Main Exclusion Criteria:

Patients who meet any of the criteria listed below will not be eligible for participation in this study. A patient will not be eligible for study participation if:

* is unable or unwilling to swallow pyrotinib;
* has been < 2 weeks since the last radiotherapy, chemotherapy, hormone therapy, surgery or molecule-target therapy (< 6 weeks if chemotherapy included nitrosoureas or mitomycin);
* the bone or skin is the only site of disease (for Part 2 extension only);
* has pleural or peritoneal only disease;
* has uncontrolled ≥ grade 2 hypokalemia and hypomagnesemia;
* has had other cancer(s) within 5 years prior to screening with the exception of contralateral breast carcinoma, adequately treated cervical carcinoma in situ, or adequately treated basal or squamous cell carcinoma of the skin;
* has active central nervous system (CNS) metastases, as indicated by clinical symptoms, cerebral edema, and/or progressive growth (patients with a history of CNS metastases or cord compression are allowable if they have been definitively treated and have been clinically stable for at least 4 weeks, and off steroids and anticonvulsants, before first dose of study drug);
* has either QTcF prolongation (> 470 ms for female and > 450 ms for male), a known history of QTcF prolongation or Torsade de Pointes; or is on drugs that are required for existing medical conditions and that may result in QT prolongation (e.g., anti-arrhythmic drugs); patients who use medications that have a minimal impact on the QTcF interval in the Arizona-CERT criteria are allowed to participate in this study at Investigator's discretion based on his/her clinical assessment);
* has a significant chronic or recent acute gastrointestinal disorder with diarrhea as a major symptom (e.g., Crohn's disease, malabsorption, or ≥ grade 2 diarrhea of any etiology at baseline);
* has participated in any other investigational drug clinical studies within the last 4 weeks;
* is concurrently receiving other anti-tumor therapies at time of study screening visit;
* has an active infection (per Investigator judgment);
* has a history of immunodeficiency including seropositive for human immunodeficiency virus, or has other acquired or congenital immunodeficient disease;
* has evidence of uncontrolled heart disease, including (1) congestive heart failure (New York Heart Association functional classification) of ≥ 2), (2) angina requiring treatment (3) myocardial infarction within the past 12 months, or (4) any clinically significant supraventricular arrhythmia or ventricular arrhythmia requiring treatment or intervention;
* has allergies or a known history of hypersensitivity to any components of the pyrotinib;
* is female and of childbearing potential (WOCBP) who is unwilling or unable to use an acceptable method (barrier methods only) to avoid pregnancy for the entire study period and for up to 28 days post last dose;
* is female and pregnant (or found to be pregnant at screening) or breastfeeding;
* evidence of significant medical illness or an abnormal laboratory finding, which according to the Investigator's judgment, will substantially increase the risk of participation in and completion of the study. Including, but not limited to, serious ongoing infection (ie, requiring intravenous antibiotic or antiviral agent), uncontrolled major seizure disorder, or significant pulmonary disorder (e.g. interstitial pneumonitis, pulmonary hypertension); hypertension (> grade 3), severe diabetes (uncontrolled > grade 3 hyperglycemia), serious ongoing infection or thyroid disease;
* has a known history of neurological psychiatric disease including epilepsy or dementia that would interfere with patient's ability to participate in the study or to provide consent;
* has had prior exposure to any other investigational HER2 targeted agents within 4 weeks of screening visit.
* is currently taking strong CYP3A4 inhibitor or concomitant meds.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2015-06; Primary Completion 2021-05 (Estimated); Study Completion 2021-06 (Estimated)

PRIMARY OUTCOMES:
Part 1 Maximum Tolerated Dose (MTD) | Day 1 to 28 ( Cycle 1)
  to assess safety and tolerability of pyrotinib with a maximum tolerated dose (MTD) of pyrotinib in patients with Human Epidermal Growth Factor Receptor 2 (HER2)-positive advanced solid tumors (metastatic breast cancer, gastric or other solid tumors with no targeted agent as standard of care).
Part 2 Overall Response Rate (ORR) | up to 24 months after the first dose
  to estimate the overall response rate (ORR) for patients with HER2-positive metastatic breast cancer (mBC) and HER2 mutant non-small cell lung cancer (NSCLC) treated at the RP2D (or MTD).

SECONDARY OUTCOMES:
Maximum plasma concentration(Cmax) | Up to 3 cycles(each cycle 28 days)
Time to Cmax | Up to 3 cycles(each cycle 28 days)
Terminal half life (t1/2) | Up to 3 cycles(each cycle 28 days)
Area under the plasma concentration-time curve | Up to 3 cycles(each cycle 28 days)
Volume of distribution(V/F) | Up to 3 cycles(each cycle 28 days)
Plasma Clearance(CL/F) | Up to 3 cycles(each cycle 28 days)
Progression Free Survival (PFS) | up to 24 months after the first dose

CONTACTS AND LOCATIONS:
Overall Officials: Junsheng Wang, MD, Study Director — Hengrui Therapeutics, Inc.
Locations (10):
- United States (10):
  - University of California, Irvine School of Medicine, Orange, California
  - UC Davis Comprehensive Cancer Center, Sacramento, California
  - Florida Cancer Specialists, Sarasota, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Henry Ford Health System, Detroit, Michigan
  - Washington University, St Louis, Missouri
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Tennessee Oncology, Nashville, Tennessee
  - South Texas Accelerated Research Therapeutics, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No